## Investigating Racial Differences in Diet Benefits for Knee Osteoarthritis

## Study Protocol & Statistical Analysis Plan

NCT04343716

08/13/2024

Robert Sorge, Associate Professor, Principal Investigator University of Alabama at Birmingham Birmingham, AL 35294

## Statistical Analysis Plan

For primary outcome measures (WOMAC pain, WOMAC function, BPI pain severity, BPI pain interference, evoked pain tests), a change score will be calculated between baseline measures and those taken at the end of the intervention. To determine whether there are differences based on racial group, an analysis of variance (ANOVA) will be carried out with "race" as the between-subjects factor. Main effects of race will be reported.

## **Revised Plan**

Following recruitment, it was determined that the limited number of non-Hispanic White (NHW) women in the study would make analysis of proposed aims impossible. Therefore, it was decided that the analysis would be altered to determine whether the non-Hispanic Black (NHB) women experienced a change over time in response to the diet intervention across the previous outcome measures. As such, all variables will be analyzed using repeated measures ANOVA and the Greenhouse-Geisser correction will be used when violations of sphericity are detected.